CLINICAL TRIAL: NCT00696891
Title: Study Comparing Immunogenicity, Reactogenicity and Safety of GSK Biologicals' HBV-MPL Vaccine With That of Engerix™-B When Both Are Injected According to 3 Dose Schedule (0, 1, 6 Months) in an Adult Population Aged Between 50 and 70 Years
Brief Title: Study Comparing Immunogenicity, Reactogenicity and Safety of GSK Bios' HBV-MPL Vaccine With That of Engerix™-B in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 208129/022
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Adjuvanted hepatitis B vaccine, hepatitis B, Engerix™-B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL vaccine
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine — 3-dose intramuscular injection
  Arms: Group A
Biological: Engerix™-B — 3-dose intramuscular injection
  Arms: Group B

SUMMARY:
This study is conducted to compare the immunogenicity, reactogenicity and safety of Engerix™-B and HBV-MPL vaccine against hepatitis B infection in an elderly population

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 to 70 years old.
* Good physical condition as established by clinical examination and history taking at the time of entry.
* Female participants who are at risk to become pregnant will be on a contraceptive programme if necessary during the study period.
* Written informed consent obtained from the subjects

Exclusion Criteria:

* Positive at screening for anti-HBV antibodies.
* Elevated serum liver enzymes
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Any chronic drug treatment, including any treatment with immunosuppressive drugs, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Simultaneous participation in any other clinical trial.
* Previous vaccination with a recombinant hepatitis B vaccine.
* Previous vaccination with an MPL containing vaccine.
* Administration of immunoglobulins in the past 6 months and during the whole study period
* Vaccination one week before and one week after each dose of the study vaccine

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 1997-06; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At Month 7

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | At Months 1, 2, 6, 7 and 12
Occurrence and intensity of solicited local symptoms | 4-day follow-up after vaccination
Occurrence and intensity and relationship to vaccination of solicited general symptoms | 4-day follow-up after vaccination
Occurrence and intensity of any symptoms (solicited/ unsolicited). | 4-day follow-up after vaccination
Occurrence, intensity and causal relationship of unsolicited symptoms | Within 30 days after vaccination
Serious adverse events | Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Clinical Trials Call Center, Wilrijk, Belgium
- GSK Clinical Trials Call Center, Toronto, Canada
- GSK Clinical Trials Call Center, Gothenburg, Sweden